CLINICAL TRIAL: NCT00118625
Title: A Double-Blind Phase IIa Study to Demonstrate the Contribution of MPL® to Tyrosine Adsorbed Birch + Hazel + Alder Pollen Allergoid (Tree MATA) With a Single-Blind Portion to Evaluate the Residual Allergenicity in Skin Test in Volunteers Allergic to Birch and Hazel and Alder Pollen
Brief Title: Assessment of the Contribution of Monophosphoryl Lipid A (MPL) to a Tree Pollen Allergy Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TreeMATAMPL202; P2DP05002
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Specific Immunotherapy; Adjuvant; Allergy Vaccination; Allergenicity
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

INTERVENTIONS:
Biological: Tree MATA MPL

SUMMARY:
Allergen-specific immunotherapy (SIT), the administration of gradually increasing quantities of an allergen extract to an allergic patient, is a curative approach which directly treats the underlying allergic disease. Tree MATA MPL has been developed to provide pre-seasonal specific immunotherapy for patients with an allergy to tree pollen (hay fever).

The tolerability and immunogenicity of Tree MATA (allergen modified with glutaraldehyde and adsorbed to tyrosine) with and without MPL adjuvant (monophosphoryl lipid A, extracted from a bacterial cell surface) is being investigated in this double-blind, randomized Phase IIa study in volunteers allergic to birch and hazel and alder pollen.

Additionally, this study will assess residual allergenicity of the modified birch and hazel and alder pollen in the product Tree MATA MPL using skin prick testing in volunteers allergic to birch and hazel and alder pollen.

DETAILED DESCRIPTION:
Allergic rhinitis is a nasal inflammatory disorder initiated by an immunoglobulin-E (IgE) mediated hypersensitivity to allergens. When a patient is exposed to an allergen to which he or she is sensitive, the allergen cross-links with the IgE antibody, which is bound to the surface of tissue mast cells. This cross-linking then triggers the release of proinflammatory substances, such as histamine and eicosanoids, and is known as the early response. In a skin prick test, this reaction produces a wheal-and-flare response. Normally, systemic exposure to an allergen also leads to the more prolonged late reaction, in which eosinophils, basophils, and activated T cells are recruited to the site of exposure. The recruited T cells also secrete inflammatory cytokines, such as interleukin-4 (IL-4) and IL-5, typically associated with helper T cells type 2 (TH2), which further propagate the inflammatory cascade. Typically, the early response occurs within 15 to 30 minutes (but as quickly as a few seconds) and usually resolves within 1 to 3 hours, and the late response occurs within 6 to 12 hours and resolves in 24 hours.

Allergic vaccination (AV), also referred to as immunotherapy or allergen-specific immunotherapy (SIT), is a curative approach that is available for allergic diseases, which directly treats the underlying disease. AV is the practice of administering gradually increasing quantities of an allergen extract to an allergic patient to ameliorate the symptoms associated with the subsequent exposure to the causative allergen. AV is believed to exert its beneficial effects on the immune system, at least in part, by modifying the T-lymphocyte response to subsequent natural allergen exposure. AV has been shown to inhibit both early and late responses to allergen exposure. AV acts on T cells to modify peripheral and mucosal TH2 responses to an allergen in favor of helper T cell type 1 (TH1) responses. One of the hallmarks of successful AV is the redressing of a "healthy" TH1/TH2-balance.

Although efficacious, immunotherapy is generally considered a long-term disease modifying measure that requires months to years of treatment, entails multiple injection regimens and involves some risk for adverse immune reactions.

Allergy Therapeutics (AT) has developed formulations over the years to increase both the safety and efficacy of such treatment. In particular, the allergen extract has been chemically modified with glutaraldehyde and formulated with L-tyrosine to act as a depot adjuvant and provide a slow release of the allergens or modified allergens. This increases the safety profile and enhances the efficacy-associated immunological changes. Efficacy could be further improved by adding the immunological adjuvant monophosphoryl lipid A (MPL).

Tree MATA MPL is designed to provide a vaccine that will be efficacious with only three escalating dose injections, in contrast to the longer schedules currently in use. It is designed to have all of the current advantages of an allergy vaccine, which can modify the underlying disease process, as opposed to pharmacological control, which treats only the symptoms. The vaccine will also be safer to use than a formulation containing a similar mass of unmodified allergen extract due to the propensity of the unmodified allergen extract to cause severe local allergic reactions or anaphylaxis, because of its reduced reactivity with IgE antibody.

The tolerability and immunogenicity of Tree MATA with and without MPL adjuvant is being investigated in this double-blind, randomized Phase IIa study in volunteers allergic to birch and hazel and alder pollen.

Additionally, this study will assess residual allergenicity of the modified birch and hazel and alder pollen in the product Tree MATA MPL using skin prick testing in volunteers allergic to birch and hazel and alder pollen.

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick test for birch and hazel and alder allergen
* Positive skin prick test to positive histamine control
* Negative skin prick test to negative control
* Specific IgE for birch as documented by a radioallergosorbent or equivalent test with class ≥ 2
* History of at least 1 season of moderate to severe seasonal rhinoconjunctivitis due to an IgE - mediated allergy to pollen from birch and hazel and alder
* Patients must score on the disease severity questionnaire as moderate or severe.
* Males or non-pregnant, non-lactating females
* Willing and able to attend required study visits
* Able to follow instructions
* Willing and able to give written informed consent

Exclusion Criteria:

* Acute or subacute atopic dermatitis and/or urticaria factitia and/or urticaria due to physical or chemical influence and/or chronic dermatitis
* Moderate to severe asthma
* Visual inspection of the forearms indicates potential problems with the conduct or interpretation of the skin prick test; both forearms must be available for testing.
* History or presence of diabetes, cancer or any clinically significant cardiac, metabolic, renal, or hematologic diseases or disorders
* Recent clinically significant history of hepatic, gastrointestinal, dermatologic, venereal, neurologic or psychiatric diseases or disorders
* Any clinically significant abnormal laboratory value at Visit 0
* Perennial allergens: clinically relevant sensitivity to house dust mites, molds and epithelia
* Patient has clinically relevant sensitivity to the following summer/autumn season flowering plants: plantain, orache, nettle, mugwort , Bermuda grass, or ragweed.
* Secondary alteration at the affected organ
* History of autoimmune diseases
* Patient is taking ß-blockers for any indication
* Patient who is not allowed to receive adrenalin
* Patients in whom tyrosine metabolism is disturbed
* Presence of a disease with a pathogenesis interfering with the immune response and patient has received medication which could influence the results of this study
* Documented evidence of acute or significant chronic infection
* History of anaphylaxis
* Documented history of angioedema
* Hypersensitivity to the excipients of the study medication
* Previous or current hyposensitization therapy with comparable tree allergen extracts
* Currently using anti-allergy medication and other drugs with antihistaminic activity
* Patients currently participating in a clinical trial or who have been exposed to study medication within the last 30 days
* Patients who cannot communicate reliably with the Investigator or who are not likely to cooperate with the requirements of the study
* Patient is pregnant or planning pregnancy and/or lactating
* Patient has received treatment with preparation containing monophosphoryl lipid A during the past 12 months
* Concurrent use of any prohibited medication(s), as listed in the study protocol.
* Any systemic disorder that could interfere with the evaluation of the study medication(s)
* Clinical history of drug or alcohol abuse, at the Investigator's discretion, that would interfere with the patient's participation in the study
* Study site staff or immediate relatives of study site staff or other individuals who would have access to the clinical study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-07; Study Completion 2005-09

PRIMARY OUTCOMES:
immunological response to Tree MATA MPL versus Tree MATA (birch specific)

SECONDARY OUTCOMES:
immunological response to Tree MATA MPL versus Tree MATA (hazel and alder specific)
allergenicity of the modified tree (birch, alder, hazel) pollen allergoid using skin prick testing
tolerability of native allergen, modified allergen and tyrosine adsorbents +/- MPL in the skin prick tests
tolerability of the different dose steps compared between Tree MATA MPL and Tree MATA treatment groups
the tolerability of the cumulative subcutaneous doses compared between Tree MATA MPL and Tree MATA treatment groups
safety laboratories
vital signs
12-lead electrocardiogram (ECG)
number of adverse events
number of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Principal Investigator — Allied Research International Inc.
Locations (1):
- Allied Research International Inc., Mississauga, Ontario, Canada